CLINICAL TRIAL: NCT00739986
Title: A Randomized, Double-Blind, Placebo-controlled Study of CNI-1493 for Treatment of Moderate to Severe Crohn's Disease 1 or 3 Days' Treatment vs. Placebo
Brief Title: Semapimod for Treatment of Moderate to Severe Crohn's Disease 1 or 3 Days' Treatment Versus Placebo
Acronym: CD04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNI-1493-CD04
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2012-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; TNF-alpha; IL-6; MAP Kinase; CNI-1493
MeSH Terms: conditions — Crohn Disease | interventions — semapimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Semapimod 60 mg IV x 1 day, placebo IV x 2 days
  Interventions: Drug: Semapimod
- 2 (Experimental): Semapimod 60 mg IV x 3 days
  Interventions: Drug: Semapimod
- 3 (Placebo Comparator): Placebo comparator IV x 3 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semapimod — semapimod 60 mg IV x 1 day, placebo x 2 days
  Arms: 1
Drug: Semapimod — Semapimod 60 mg IV x 3 days
  Arms: 2
Drug: Placebo — placebo IV x 3 days
  Arms: 3

SUMMARY:
Assessment of the number of days' treatment with semapimod necessary for efficacy, as measured by response rate to CNI-1493 as compared to placebo, in patients with moderate to severe Crohn's disease (CD).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women at least 18 years of age.
2. Baseline Crohn's Disease Activity Index (CDAI) 250-400.
3. Crohn's disease of at least 3 months duration, with colitis, ileitis, or ileocolitis, confirmed by radiography and/or endoscopy.
4. Those of childbearing potential were to use a barrier method (diaphragm or condom) of contraception and continue doing so for at least 3 months after last study medication. It was recommended that two forms be used.
5. Patients receiving medications for CD were to be on each medication for at least 8 weeks prior to screening and on stable doses of each for at least 2 weeks prior to screening, with the following exceptions:

   * those on methotrexate had to be on a stable dose for at least 4 weeks and not be receiving more than 25 mg/wk
   * those on azathioprine or 6-mercaptopurine on a stable dose for at least 10 weeks
   * those on steroids had to have been on steroids for at least 2 weeks and on a stable dose for those 2 weeks. They were not to be receiving more than 20 mg/day prednisone or equivalent
   * those on mesalazine had to have been on for at least 6 weeks and on a stable dose for at least 2 weeks
   * those on antibiotics for CD had to have been on for at least 2 weeks and on a stable dose for those 2 weeks
6. Any CD medication which had been discontinued was to have been discontinued at least 4 weeks prior to screening, with the exception of infliximab, which was to have been discontinued at least 8 weeks prior to screening.
7. The screening laboratory tests were to meet the following criteria:

   Hgb >= 8.5 g/dL (5.3 mmol/L) WBC 3.5-20 x 109/L Neutrophils >= 1.5 x 109/L Platelets >= 100 x 109/L ALT (SGPT) <1.5 x the upper limit of normal range Alkaline phosphatase <2.5 x the upper limit of normal range Bilirubin <25 mmol/L (1.5 mg/dl) Creatinine <110 mol/L (1.2 mg/dl)
8. Patients were to be able to adhere to the study visit schedule and/or protocol requirements.
9. Patients were to be able to give informed consent and the consent was to be obtained prior to any study specific screening procedures.

Exclusion Criteria:

1. Treatment with any other experimental therapeutics within the last 4 weeks before enrolment.
2. History of tuberculosis, either clinically or as evidenced by a positive chest x-ray (exclusion criterion #8) or PPD.
3. Patients who had received anti-TNF therapy, such as infliximab, within 8 weeks of screening for this study. Patients who had received anti-TNF therapy >8 weeks prior to screening were eligible.
4. Patients with any ostomy, extensive bowel resection (e.g., more than 100cm of small bowel, proctocolectomy or colectomy with ileorectal anastomosis). Segmental colectomy was permitted.
5. Patients immediately in need of surgery for active gastrointestinal bleeding, peritonitis, intestinal obstruction, or intra-abdominal or pancreatic abscess requiring surgical drainage.
6. Patients with known severe fixed symptomatic stenosis of the small or large intestine.
7. Evidence at the time of enrolment of bowel obstruction or history within the preceding six months as confirmed by radiography, endoscopy, or surgery.
8. Patients with a clinically significant abnormality or granulomata or any other evidence of primary tuberculosis infection on chest X-ray
9. Patients with current signs or symptoms of clinically significant hematologic, endocrine, pulmonary, cardiac, neurologic or cerebral disease.
10. Patients with previous diagnosis of, or known, malignancies.
11. Patients with serious infections, such as hepatitis, HIV, pneumonia or pyelonephritis, within 3 months prior to screening.
12. History of opportunistic infections such as herpes zoster within 2 months prior to screening, evidence of active CMV, active Pneumocystis carinii, drug resistant atypical mycobacterium.
13. Patients with stool examination positive for enteric pathogens, pathogenic ova or parasites, or Clostridium difficile toxin.
14. Women who were pregnant or breast-feeding.
15. A psychiatric, addictive, or any disorder that compromises ability to give truly informed consent for participation in this study.
16. Patients who had received CNI-1493 in the past.
17. More than three doses of NSAIDs, including aspirin and COX-2 inhibitors, within the two weeks prior to start of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2002-10; Primary Completion 2004-06 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Crohn's Disease Activity Index (CDAI) score | Day 29

SECONDARY OUTCOMES:
Inflammatory Bowel Disease Questionnaire (IBDQ) | Day 29
Crohn's disease endoscopic index of severity (CDEIS) | Day 29
Change in level of C-reactive protein (CRP) | Day 29
Safety (Adverse events) | Days 29 and 57

CONTACTS AND LOCATIONS:
Overall Officials: Daan Hommes, MD, Principal Investigator — Academic Medical Center, Netherlands
Locations (28):
- United States (10):
  - Institute of Healthcare Assessment, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Advanced Gastroenterology Associates, Suwanee, Georgia
  - Northwestern University, Chicago, Illinois
  - Long Island Clinical Research Associates, Great Neck, New York
  - Asher Kornbluth, MD, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Gastroenterology Associates, Bristol, Tennessee
  - Gastroenterology Associates, Kingsport, Tennessee
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Academic Hospital Gasthuisberg, Leuven
- Germany (7):
  - Benjamin Franklin University, Berlin
  - Medizinischen Hochschule-Hannover, Hanover
  - Universitats Klinikum Heidelberg, Heidelberg
  - University of Kiel, Kiel
  - Gastroenterologische Fachpraxis, Minden
  - Stadtisches Krankenhaus Munchen-Bogenhausen, München
  - University of Munster, Münster
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Shaare Zedek Hospital, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Netherlands (4):
  - Academic Medical Center, Amsterdam
  - Free University (Vrije Universiteit), Amsterdam
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Erasmus Medical Center, Rotterdam